

9 February 2021

## Consent form

| I amfreely and voluntary consent to participate in research study under the direction of researcher / Mohamed Hesham Sayed and |
|---|
| Samah Mahmoud Sheha. |
| A thorough description of the procedures has explained, and I understand that I may withdraw my consent and discontinue participation in this research at any time without prejudice to me. |
| Date Participant |